CLINICAL TRIAL: NCT02362737
Title: Active and Healthy Brotherhood: A Program for Chronic Disease Self-Management for Black Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gramercy Research Group (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Arizona State University (Other); Project Brotherhood (Unknown); University of North Carolina, Chapel Hill (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AD-1403-11098
Record Dates: First submitted 2015-01-30; First posted 2015-02-13 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Chronic Disease; Obesity; Hypertension; Diabetes; Self Care; Medication Adherence
MeSH Terms: conditions — Chronic Disease; Obesity; Hypertension; Diabetes Mellitus; Medication Adherence | interventions — Exercise

ARMS (2):
- Active and Healthy Brotherhood (AHB) (Experimental): 16-week behavioral intervention
  Interventions: Behavioral: Active and Healthy Brotherhood (AHB)
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Active and Healthy Brotherhood (AHB) — Participants will attend group sessions led by trained group facilitators. The group sessions will be ~16 weekly meetings of ~90 minutes duration for 4 months. AHB participants will also engage in experiential learning opportunities. Following the intensive intervention phase, during months 5 and 6, participants will receive three structured, individual phone calls with the group facilitator.
  Arms: Active and Healthy Brotherhood (AHB)

SUMMARY:
This study will test ways to improve health behaviors using an intervention that has been specially designed for African-American men. The program, called Active & Healthy Brotherhood (AHB), will provide information on basic health, and healthy eating, physical activity, stress management, and how to get medical care when needed.The AHB intervention will be compared to a control group that will receive basic health information in videos and brochures.

ELIGIBILITY:
Inclusion Criteria:

1. AA (based on self-report)
2. self-reported male
3. aged at least 21 years
4. non-institutionalized (i.e., community-dwelling, not living in assisted living facilities, nursing homes, etc.)
5. at high risk for developing chronic disease (e.g., not meeting current guidelines for PA and/or F&V intake; current smoker; diagnosed with high cholesterol) or
6. currently diagnosed with diabetes, hypertension, or cardiovascular disease
7. residents of Forsyth County, NC (or surrounding areas and able to attend group sessions in Forsyth County).

Exclusion Criteria:

1. have had a cardiovascular procedure (e.g., heart surgery), heart attack, heart failure, stroke in the last 6 months
2. have cognitive, visual, auditory, physical functional (e.g., unable to walk unassisted), or language impairment precluding participation in group discussion, learning activities, or data collection.
3. currently achieve >150 min/wk of moderate intensity PA or >75 min/wk of vigorous intensity PA AND currently consume > 9 servings of F&V daily.
4. are currently enrolled in a chronic disease management program.
5. are unwilling to accept randomization assignment or planning to move from local area in <2 years.
6. are currently receiving chemotherapy/radiation treatments.

Participants will be required to obtain approval from a health care provider prior to participation in the study if they:

1. are unable to participate in moderate PA due to physical limitations as indicated by positive (risk) responses on the PA Readiness Questionnaire (PAR-Q) and/or physician disapproval on the PAR Medical Examination.
2. have BP>180/>110 and/or HbA1C>12 and/or triglycerides >500.
3. have health conditions that could preclude changes to diet (e.g., irritable bowel syndrome, celiac disease)

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 332 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change activity behavior (minutes per week in Total physical activity (PA) and light, moderate, vigorous PA). | baseline, 6 months, 12 months
  Minutes per week in Total physical activity (PA) and light, moderate, vigorous PA
Change sedentary behavior (minutes per week of sedentary behavior). | baseline, 6 months, 12 months
  Minutes per week of sedentary behavior
Change dietary intake (Fruit and vegetable servings, % fat, sodium and fiber intake). | baseline, 6 months, 12 months
  Fruit and vegetable servings, % fat, sodium and fiber intake
Change stress management. | baseline, 6 months, 12 months
  Identification of issues and strategies that affect stress management
Change help-seeking behaviors (Medication adherence and doctor/ER visits). | baseline, 6 months, 12 months
  Medication adherence and doctor/ER visits

SECONDARY OUTCOMES:
Change blood pressure. | baseline, 6 months, 12 months
Change body weight. | baseline, 6 months, 12 months
Change blood glucose. | baseline, 6 months, 12 months
Change HbA1c. | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gramercy Research Group, Winston-Salem, North Carolina, United States